CLINICAL TRIAL: NCT03793283
Title: Effectiveness and Safety of Continuous Subcutaneous Insulin Infusion Versus Multiple Dose Insulin Injections in Type 1 Diabetes Mellitus Adult Patients in Routine Clinical Practice
Brief Title: Continuous Subcutaneous Insulin Infusion Versus Multiple Dose Insulin Injections in Routine Clinical Practice
Acronym: real-ECIMI
Status: Completed | Type: Observational
Sponsor: Castilla-La Mancha Health Service (Other)
Collaborators: University of Castilla-La Mancha (Other); Universidad de Córdoba (Other)
Responsible Party: Principal Investigator, Jesús Moreno Fernández, Principal investigator, Castilla-La Mancha Health Service
Other Study IDs: C-225
Record Dates: First submitted 2018-12-27; First posted 2019-01-04 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Continous Subcutaneous Insulin Infusion: All T1DM adult patients attended in Ciudad Real General University Hospital and treated with CSII.
  Forty-five patients are actually treated with CSII in our hospital.
  Interventions: Device: CSII
- Multiple dose insulin injections (MDI):: Forty-five T1DM adult patients attended in Ciudad Real General University Hospital and treated with MDI.
  MDI patients will be selected through simple random sampling (1:1) from our T1DM patient database.
  Interventions: Drug: Multiple dose insulin injections

INTERVENTIONS:
Device: CSII — Currently receiving CSII therapy during 6 or more months.
  Other Names: Continuous subcutaneous insulin infusion
  Groups: Continous Subcutaneous Insulin Infusion
Drug: Multiple dose insulin injections — Currently receiving MDI therapy during 6 or more months.
  Other Names: MDI
  Groups: Multiple dose insulin injections (MDI):

SUMMARY:
Observational study about effectiveness and safety of continuous subcutaneous insulin infusion compared to multiple dose insulin injections in Type 1 Diabetes Mellitus (T1DM) adult patients in routine clinical practice.

DETAILED DESCRIPTION:
Cross-sectional analysis about effectiveness and safety of continuous subcutaneous insulin infusion compared to multiple dose insulin injections in T1DM adult patients in routine clinical practice.

All clinical variables are gathered from four EMR softwares (Mambrino XXI, Carelink Pro®, Emminens eConecta® and FreeStyle Libre®).

Data analysis is conducted using SPSS (Chicago, IL) statistics software. Results are presented as mean ± SD values or percentages. A paired Student's t-test or a Wilcoxon signed-rank test were used for the analysis of differences. Comparisons between proportions were analyzed using a chi-squared test. A P value < 0.05 was considered statistically significant.

The protocol was approved by the reference Castilla-La Mancha Public Health Institute Ethic Committee. All participants provided written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age.
* Diagnosed of Type 1 Diabetes Mellitus.
* Be attended in Ciudad Real General University Hospital.
* Current treated with CSII (CSII cohort) or MDI (MDI cohort) during ≥6 months.

Exclusion Criteria:

* Less than 18 years old.
* Other types of diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Forty-five T1DM adult patients attended in Ciudad Real General University Hospital and treated with CSII.
  MDI patients will be selected through simple random sampling (1:1) from our T1DM patient database.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Concentration of Hemoglobin A1C (HbA1C). | 1 year
  Between group hemoglobin A1C (HbA1C) difference. Physiological parameter. Unit of measure: %.

SECONDARY OUTCOMES:
Hypoglycemia frequency. | 1 year
  Between group hypoglycemic frequency difference. Unit of measure: daily number of events of glycemic values <70 mg/dL.
Concentration of Capillary blood glucose. | 1 year
  Between group capillary blood glucose difference. Physiological parameter. Unit of measure: mg/dL.
Concentration of Interstitial blood glucose. | 1 year
  Between group interstitial blood glucose difference. Physiological parameter. Unit of measure: mg/dL.
Glycemic variability: coefficient of variation of capilary/interstitial blood glucose. | 1 year
  Glycemic variability expressed as coefficient of variation of capilary/interstitial blood glucose.
  Physiological parameter. Unit of measure: %.
Glycemic variability: standar deviation of capilary/interstitial blood glucose. | 1 year
  Glycemic variability expressed as standar deviation of capilary/interstitial blood glucose.
  Physiological parameter. Unit of measure: mg/dL.
Self-monitoring of blood glucose (SMBG) daily frequency | 1 year
  Self-monitoring of blood glucose (SMBG) daily frequency. Unit of measure: number of daily controls.
Severe hypoglycemia frequency. | 1 year
  Number of events during the last year of severe hypoglycemia frequency defined as any glycemic value <70 mg/dL requiring assitance from another person to treat.
  Unit of measure: number of events during the last 12 months.
Weight. | 1 year
  Between group weight differences. Physiological parameter. Unit of measure: Kg.
Insuline dose. | 1 year
  Daily insulin doses (basal and bolus) and bolus insulin daily frequency. Unit of measure: IU/Kg/24h.
Diabetes quality of life (DQOL). | 1 year.
  Diabetes related quality of life (EsDQOL questionnary). Spanihs version of DQOL questionnary. Unit of measure: Questionnary score. Higher values represent a worse outcome. Forty-six questions in four categories: Satisfaction (15), Impact (20), Social/vacational worryness (7) and Diabetes related worryness (4). Each question score from 1 to 5 points.
  Total minimum score 46, total maximum score 230. Satisfaction range from 15 to 75, Impact range from 20 to 100, Social/vacational worryness range from 7 to 35 and Diabetes related worryness range from 4 to 20.
Satisfaction with the treatment received: Diabetes Treatment Satisfaction Questionnaire Stable | 1 year
  Satisfaction with the treatment received (Diabetes Treatment Satisfaction Questionnaire Stable, EsDTSQs questionnary).
  Spanish version of DTSQs questionnary. Unit of measure: Questionnary score. Higher values represent a better outcome. Eight questions with seven possible answers ranged each one from 0 to 6 points. First six questions compute a subscore ranged from 0 to 36 points. Two last questions are independtly analyzed (each one range from 0 to 6 points).
Unawareness hypoglycemia. | 1 year.
  Unawareness hypoglycemia frequency (Clarke questionnary). Unit of measure: Questionnary score. Higher values represent a worse outcome. Eight questions with each answer categorized in normal (A) or abnormal (R). Total sum of abnormal (R) answers classifed patients in normal perception (range from 0 to 2), indeterminate percepction (range=3) and abnormal perception (range from 4 to 8).
Safety related adverse events. | 1 year
  Serious related adverse events: diabetes ketoacidosis, hospitalization, death. Unit of measure: number of events.

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Moreno-Fernandez, PhD, Principal Investigator — Castilla-La Mancha Public Health Service.
Locations (1):
- Obispo Rafael Torija, St., Ciudad Real, Spain

IPD SHARING:
Plan to Share IPD: No